CLINICAL TRIAL: NCT04838379
Title: Perioperative Analgesic Effect of Preemptive Ultrasound Guided Rectus Sheath Block and Transversus Abdominis Plane Block With Dexmedetomidine vs Dexamethasone for Laparoscopic Surgery in Paediatrics
Brief Title: Ultrasound Guided Rectus Sheath Block and Transversus Abdominis Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kirolos Gamal Reda, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01210861577
Record Dates: First submitted 2021-03-31; First posted 2021-04-09 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Cholecystitis; Appendicitis
Keywords: us guided rectus sheath block&tap block; laparscopic surgery; regional anesthesia
MeSH Terms: conditions — Cholecystitis; Appendicitis | interventions — Dexmedetomidine; Dexamethasone; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Age: 8-12years.
  * Weight: 20-60 kg.
  * Sex: both males and females.
  * ASA physical status: I-II.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group Bupivacaine (Placebo Comparator): will include 30 patients: each one will receive 2.5 mg/kg of 0.25% bupivacaine diluted in a 20 mL syringe of normal saline, 10 minutes before skin incision
  Interventions: Drug: Dexmedetomidine
- group bupivacaine&dex (Active Comparator): will include 30 patients: each one will receive 2.5mg/kg of 0.25% bupivacaine plus 1 µ/kg of dexmedetomidine diluted in a 20 mL syringe of normal saline, 10 minutes before skin incision
  Interventions: Drug: Dexmedetomidine
- Group bupivacaine & dexamethasone (Active Comparator): will include 30 patients: each one will receive 2.5 mg/kg of 0.25% bupivacaine plus dexamethasone (0.3 mg/kg) diluted in a 20 mL syringe of normal saline , 10 minutes before skin incision
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Ninety patients were randomized to receive ultrasound-guided RSB&tap block After the induction of anesthesia and patient stabilization, the abdomen was sterilized and draped. Then, under complete aseptic conditions, ultrasound-guided Bilateral Rectus Sheath Block & tap block was performed
  Other Names: Dexamethasone; Bupivacaine

SUMMARY:
The current study aimed to assess the efficacy of Dexmedetomidine (DEX) and Dexamethasone as an adjuvant to ultrasound guided TAP and RS block to prolongation of postoperative analgesia and better pain control in children undergoing laparoscopic surgeries

DETAILED DESCRIPTION:
Laparoscopic surgeries are one of the most frequently performed paediatric surgeries . Although minimally invasive, this technique is still associated with a significant amount of pain and anxiety in children . Indeed, children who are highly anxious prior to surgery tend to have more postoperative pain, delayed hospital discharge, and higher incidence of emergence delirium, sleep disturbances, and other mal-adaptive behaviour changes that can last up to a few weeks following surgery . To improve analgesia and decrease postoperative anxiety in children undergoing laparoscopic appendectomies multimodal approach for pain control can be employed.

Over the past years, the concept of pain management has extended from simply decreasing pain intensity to optimizing patient's condition. The goal is to decrease pain scores, stress response that should be avoided in patients, particularly cardiac patients, together with a decrease in analgesics-related adverse effects like nausea, vomiting, retention of urine and over sedation. By achieving these goals, we can certainly facilitate patient recovery and minimize the hospital stay. Improved pain control can be achieved by a combination of different types of regional analgesia with systemic analgesics. The main contributor to pain post abdominal operations is the pain from abdominal wall incision .

Many procedures were followed to decrease this intense postoperative pain such as, epidural catheter analgesia, transversus abdominis plane (TAP) block, local wound infiltration, Patient-Controlled Analgesia (PCA), peripheral nerve blocks, in addition to systemic administration of Non-Steroidal Anti- Inflammatory Drugs (NSAIDs) or opioids .

The transversus abdominis plane (TAP) block is a regional anesthetic technique that provides analgesia to the parietal peritoneum as well as to the skin and muscles of the anterior abdominal wall (9-10). Despite a relatively low risk of complications and a high success rate using modern techniques, TAP block remains overwhelmingly underused. Although the technique is technically straightforward, it has not been adopted in clinical practice .

Moreover, The Rectus Sheath Block (RSB) is one of these regional techniques that are suitable for operations with a midline incision or laparoscopic surgery with the main incision at the umbilical port. A previous study showed the analgesic efficacy of ultrasound guided rectus sheath block for laparoscopic appendectomy compared to a control group injected with saline instead of a local anesthetic Generally, in laparoscopic surgeries, the sites of port incision are associated with considerable postoperative discomfort. Thus, we performed TAP and RS block to ameliorate postoperative pain and improve patient outcomes. In addition to the usefulness of traditional local anesthetics to provide analgesia during the course of the postoperative period is restricted by their short duration of action .

Dexmedetomidine (DEX) and Dexamethasone has been shown as a valuable additives to local anesthetics in neuraxial blocks and peripheral nerve blocks leading to prolongation of postoperative analgesia and better pain control .

Dexmedetomidine (DEX) α-2 adrenergic receptor consists of three α-2 isoreceptors (α-2a, α-2b and α-2c), which regulate the various pharmacodynamic effects of this drug . The α-2a receptor seems to promote sedation and anxiolysis in the locus coeruleus, as well as to generate bradycardia and peripheral vasodilation by stimulation of the cerebral vasomotor center. The α-2b receptor prevents tremor, generates analgesia in the dorsal horns of the spinal cord and determines peripheral vasoconstriction. The α-2c receptor modulates the mental state .

Dexamethasone, a high-potency, long-acting glucocorticoid, has been shown to prolong peripheral nerve blockade . Dexamethasone binds to glucocorticoid receptors and inhibits potassium conductance, which decreases nociceptive C-fiber activity . Dexamethasone may also extend the duration of analgesia via local vasoconstrictive and systemic anti-inflammatory effects .

Thus, we performed TAP and RS block to ameliorate postoperative pain and improve patient outcomes.

.

ELIGIBILITY:
Inclusion Criteria:

* ● Age: 8-12years.

  * Weight: 20-60 kg.
  * Sex: both males and females.
  * ASA physical status: I-II.

Exclusion Criteria:

* • Patient's guardian refusal to participate in the study.

  * Patients having known hypersensitivity to dexametomidine will be excluded.
  * Patients with cardiovascular, liver or renal disease, unsatisfactory preoperative peripheral arterial oxygen saturation, neurological or psychiatric disease and coagulation disturbances.
  * Any perioperative cardiovascular or respiratory event occurred or difficulties in pain perception and assessment which make the study intervention clinically unacceptable.
  * Patients on regular use of analgesic or who received analgesic 24 h before surgery

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
evaluate the first call for rescue analgesia | 24 hours after recovery from anesthesia
  the time of the first call for analgesia is recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt